CLINICAL TRIAL: NCT04843059
Title: ERASE VITILIGO Early Repigmentation Approach for Stopping the Evolution of VITILIGO Prospective Multicentric Interventional Study With Blinded Evaluation
Acronym: ERASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21-PP-01
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: To compare the resident memory T-cell infiltrate in perilesional vitiligo skin after 6 months of treatment with OMP and UVB, between three groups of patients suffering from non-segmental vitiligo, using flow cytometric analysis.
  * First group will include patients with a long-lasting disease (more than 2 years) and no new or growing lesions for at least 2 years: Old vitiligo with Old lesions
  * The second group will include patients with a long-lasting disease (more than 2 years) and with at least one new lesion developed in the last 6 months: Old vitiligo with new lesions
  * The third one will include patients developing, for the first-time, vitiligo lesions with all the lesions no older than 6 months: New vitiligo
Masking Description: To compare the resident memory T-cell infiltrate in perilesional vitiligo skin after 6 months of treatment with OMP and UVB, between three groups of patients suffering from non-segmental vitiligo, using flow cytometric analysis.
  * First group will include patients with a long-lasting disease (more than 2 years) and no new or growing lesions for at least 2 years: Old vitiligo with Old lesions
  * The second group will include patients with a long-lasting disease (more than 2 years) and with at least one new lesion developed in the last 6 months: Old vitiligo with new lesions
  * The third one will include patients developing, for the first-time, vitiligo lesions with all the lesions no older than 6 months: New vitiligo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the resident memory T-cell infiltrate in perilesional vitiligo skin (Other): To compare the resident memory T-cell infiltrate in perilesional vitiligo skin after 6 months of treatment with OMP and UVB, between three groups of patients suffering from non-segmental vitiligo, using flow cytometric analysis.
  * First group will include patients with a long-lasting disease (more than 2 years) and no new or growing lesions for at least 2 years: Old vitiligo with Old lesions
  * The second group will include patients with a long-lasting disease (more than 2 years) and with at least one new lesion developed in the last 6 months: Old vitiligo with new lesions
  * The third one will include patients developing, for the first-time, vitiligo lesions with all the lesions no older than 6 months: New vitiligo
  Interventions: Other: The resident memory T-cell infiltrate in perilesional vitiligo skin

INTERVENTIONS:
Other: The resident memory T-cell infiltrate in perilesional vitiligo skin — The 3 groups will receive a combination of narrowband UVB (Nb-UVB) 3 times a week and oral mini pulses of systemic steroids (5 mg of d medrol 16mg twice a week) for 24 weeks.
  Three visits will be done (inclusion, Week 12 and 24) A skin biopsy will be done on lesional and peri-lesional area at baseline. Another skin biopsy will be taken after 24 weeks but only in perilesional area. A blood sample for assessing the circulating memory T cells and for checking the tolerance will be performed at baseline, then at W12 and W24.

SUMMARY:
Vitiligo affects 1 to 2% of worldwide population and has a demonstrated impact on the quality of life.

Optimal treatment of vitiligo requires to target the auto-immune inflammatory response (to halt the depigmentation process), in particular T cells, but also to induce the differentiation of melanocyte stem cells (to induce repigmentation). Ultimately, the treatment should also prevent the recurrences of depigmentation. Indeed, when repigmentation is achieved, 40 to 50% of lesions reoccur within one year, suggesting that skin resident memory T cell clones remain in repigmented vitiligo skin and might explain these recurrences.

The investigators hypothesize that a very early intervention could prevent the accumulation of the skin resident memory T cells in vitiligo lesions. Moreover, they also think that such an early treatment would also optimize the repigmentation process, even in traditionally resistant areas, as some remaining pre-melanocytes and maybe even some melanocytes, could proliferate and recolonize the epidermis.

Objectives : to compare the resident memory T-cell infiltrate in perilesional vitiligo skin after 6 months of treatment with OMP and UVB, between three groups of patients suffering from non-segmental vitiligo Interventions The 3 groups will receive a combination of narrowband UVB (Nb-UVB) 3 times a week and oral mini pulses of systemic steroids (5 mg of d medrol 16mg twice a week) for 24 weeks.

Three visits will be done (inclusion, Week 12 and 24) A skin biopsy will be done on lesional and peri-lesional area at baseline. Another skin biopsy will be taken after 24 weeks but only in perilesional area. A blood sample for assessing the circulating memory T cells and for checking the tolerance will be performed at baseline, then at W12 and W24.

The combination of narrowband UVB and oral minipulse of steroids are considered as a standard care of active vitiligo patients. Clinical assessment (including blood pressure) and hemogram, liver enzymes, urea, creatinemia, glycemia, natremia and kaliema will be assessed at baseline, 3 and 6 months.

Main criteria of evaluation:

The target lesion will be chosen before any treatment. The minimal size will be 2cm². Considering that skin on the face usually responds very well whilst that of hands and feet respond poorly, to avoid potential bias due to the location of treatment, these locations won't be taken as target lesions. In any cases, no biopsy will be taken on the face or in the folds.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with non-segmental vitiligo. 3 groups of patients will be selected:
* Patients with a long-lasting disease (more than 2 years) and no new or growing lesion since at least 2 years
* Patients with a long-lasting disease (more than 2 years) and with at least one new lesion since less than 6 months
* Patients developing for the first-time vitiligo lesions with all the lesions no older than 6 months 2. ≥ 18 and <35 years to have a homogeneous distribution of age between the three groups, as 80% of vitiligo cases start before the age of 30.

  3. Patient with at least one lesion of more than 2 cm² not located on the face, hands or feet.

  4. Patient needing a treatment with oral minipulses of steroids and phototherapy 5. For women of child-bearing age, an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study. A urine pregnancy test (βHCG in urines) will be performed.

  6. Affiliation to a social security system 7. Signed informed consent

Exclusion Criteria:

* 1. Pregnant or breast-feeding women. Or women who plan to get pregnant during the study duration.

  2. Segmental or mixed vitiligo 3. Vitiligo located only on face, hands and feet 4. Exposure to solar or artificial UV during the months before inclusion 5. Concomitant use of topical or systemic immunosuppressive medication or steroids 6. Patients suffering from photodermatosis or taking photosensitive drugs 7. Personal history of skin cancer. 8. Patients with diabetes, high blood pressure, osteoporosis or any other contra-indication to the use of systemic steroids.

  9. Vulnerable people: pregnant or breast-feeding women, minors, adult under guardianship or deprived of freedom 10. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
The percentage of resident memory T-cells (ratio memory T cells (CD4+CD69++ and CD8+CD69+)/Total CD4+ and CD8+ *100), assessed by cytometric analysis, in the perilesional skin of the target lesion. | at 6 months
  The target lesion will be chosen before any treatment. The minimal size will be 2cm². Considering that skin on the face usually responds very well whilst that of hands and feet respond poorly, to avoid potential bias due to the location of treatment, these locations won't be taken as target lesions. In any cases, no biopsy will be taken on the face or in the folds.

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (2):
- France (2):
  - CHU de Nice, Nice, alpes maritimes
  - CHU Bordeaux, Bordeaux

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marin Dit Bertoud Q, Bertold C, Ezzedine K, Pandya AG, Cherel M, Castillo Martinez A, Seguy MA, Abdallah M, Bae JM, Bohm M, Parsad D, Rosmarin D, Wolkerstorfer A, Bahadoran P, Blaise M, Dugourd PM, Philippo V, Delaval JM, Passeron T. Reliability and agreement testing of a new automated measurement method to determine facial vitiligo extent using standardized ultraviolet images and a dedicated algorithm. Br J Dermatol. 2023 Dec 20;190(1):62-69. doi: 10.1093/bjd/ljad304. PMID 37615581